CLINICAL TRIAL: NCT05203497
Title: SPECT Imaging of Human Epidermal Growth Factor Receptor 2 (HER2) Expression in Breast Cancer Using Technetium-99m-labelled Affibody Molecule-based Tracer 99mTc-ZHER2:41071.
Brief Title: Molecular Imaging of HER2 Expression in Breast Cancer Using 99mTc-ZHER2.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 99mTc-ZHER2
Record Dates: First submitted 2021-12-30; First posted 2022-01-24 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer Female
Keywords: 99mTc-ZHER2:41071; Breast Cancer; HER2 expression
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The tested injected doses of 99mTc-ZHER2:41071 500 μg (Experimental): At least five (5) evaluable subjects with HER2-positive status and at least five (5) subjects with HER2-negative status have to be enrolled in the study for each tested protein dose.
  Subjects withdrawn from the study for any reason will be replaced.
  Interventions: Drug: SPECT
- The tested injected doses of 99mTc-ZHER2:41071 1000 μg (Experimental): At least five (5) evaluable subjects with HER2-positive status and at least five (5) subjects with HER2-negative status have to be enrolled in the study for each tested protein dose.
  Subjects withdrawn from the study for any reason will be replaced.
  Interventions: Drug: SPECT

INTERVENTIONS:
Drug: SPECT — One single injection of 99mTc-ZHER2:41071, followed by gamma camera imaging after 2, 4, 6 and 24 hours.
  Other Names: 99mTc-ZHER2:41071

SUMMARY:
The study should evaluate distribution of 99mTc-ZHER2:41071 Affibody molecule in patients with primary HER2-positive and HER2-negative breast cancer

The primary objectives are:

1. To assess distribution of 99mTc-ZHER2:41071 in normal tissues and in tumors over time;
2. To evaluate dosimetry of 99mTc-ZHER2:41071;
3. To obtain initial information concerning safety and tolerability of 99mTc-ZHER2:41071 after single intravenous injection:

The secondary objectives are:

1. To compare the tumor imaging data with the data concerning HER2 expression obtained by immunohistochemistry (IHC) and/or fluorescent in situ hybridization (FISH) analysis of biopsy samples.

DETAILED DESCRIPTION:
Overall goal of the project: To determine HER2 expression level in primary breast cancer and possibly in axillary lymph node metastases before neoadjuvant targeted (trastuzumab or trastuzumab+pertuzumab) therapy.

Phase I. Distribution of 99mTc-ZHER2:41071 in patients with primary breast cancer.

The study should evaluate distribution of 99mTc-ZHER2:41071 in patients with primary HER2-positive and HER2-negative breast cancer.

The primary objectives are:

1. To assess distribution of 99mTc-ZHER2:41071 in normal tissues and in tumors over time;
2. To evaluate dosimetry of 99mTc-ZHER2:41071;
3. To obtain initial information concerning safety and tolerability of 99mTc-ZHER2:41071 after single intravenous injection:

The secondary objectives are:

1. To compare the tumour imaging data with the concerning HER2 expression obtained by immunohistochemistry (IHC) or fluorescent in situ hybridization (FISH) analysis of biopsy samples:

Methodology:

Open-label, exploratory, single center study. The subjects will receive a single injection of the labelled tracer.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is > 18 years of age
2. Diagnosis of primary breast cancer with possible lymph node metastases
3. Availability of results from HER2 status previously determined on material from the primary tumor, either

   1. HER2-positive, defined as a DAKO HercepTest™ score of 3+ or FISH positive or
   2. HER2-negative, defined as a DAKO HercepTest™ score of 0 or 1+; or else if 2+ then FISH negative
4. Volumetrically quantifiable tumour lesions on CT or MRI, with at least one lesion > 2.0 cm in greatest diameter outside of the liver and kidneys
5. Hematological, liver and renal function test results within the following limits:

   * White blood cell count: > 2.0 x 109/L
   * Hemoglobin: > 80 g/L
   * Platelets: > 50.0 x 109/L
   * ALT, ALP, AST: =< 5.0 times Upper Limit of Normal
   * Bilirubin =< 2.0 times Upper Limit of Normal
   * Serum creatinine: Within Normal Limits
6. A negative pregnancy test for all patients of childbearing potential. Sexually active women of childbearing potential participating in the study must use a medically acceptable form of contraception for at least 30 days after study termination
7. Subject is capable to undergo the diagnostic investigations to be performed in the study
8. Informed consent

Exclusion Criteria:

1. Second, non-breast malignancy
2. Active current autoimmune disease or history of autoimmune disease
3. Active infection or history of severe infection within the previous 3 months (if clinically relevant at screening)
4. Known HIV positive or chronically active hepatitis B or C
5. Administration of other investigational medicinal product within 30 days of screening
6. Ongoing toxicity > grade 2 from previous standard or investigational therapies, according to US National Cancer Institute's

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with primary breast cancer
Enrollment: 30 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Gamma camera-based whole-body 99mTc-ZHER2:41071 uptake value (% per organ) | 24 hours
  Whole-body 99mTc-ZHER2:41071 uptake coinciding with normal organs and tissues will be assessed using gamma camera at 2, 4, 6 and 24 hours after injection and calculated as percentage (%) of the injected dose of the radiopharmaceutical
SPECT/CT-based 99mTc-ZHER2:41071 uptake value in tumor lesions (kcounts)/SUV | 6 hours
  99mTc-ZHER2:41071 focal uptake coinciding with tumor lesions will be assessed using SPECT/CT at 2, 4 and 6 hours after injection and measured in kcounts and SUV
SPECT-based 99mTc-ZHER2:41071 background uptake value (kcounts)/SUV | 6 hours
  Uptake of 99mTc-ZHER2:41071 in the regions without pathological findings will be assessed using SPECT/CT at 2, 4 and 6 hours after injection and measured in kcounts and SUV.
Tumor-to-background ratio (SPECT) | 6 hours
  The SPECT-based tumor-to-background ratio will be calculated as follows: the value of 99mTc-ZHER2:41071 uptake coinciding with tumor lesions (kcounts) will be divided by the value of 99mTc-ZHER2:41071 uptake coinciding with the regions without pathological findings (kcounts)

SECONDARY OUTCOMES:
Safety attributable to 99mTc-ZHER2:41071 injections (physical examination) | 24 hours
  The safety attributable to 99mTc-ZHER2:41071 injections will be evaluated based on the assessments of physical examination (% of cases with abnormal findings relative to baseline)
Safety attributable to 99mTc-ZHER2:41071 injections (vital signs) | 24 hours
  The safety attributable to 99mTc-ZHER2:41071 injections will be evaluated based on the assessments of vital signs (% of cases with abnormal findings relative to baseline)
Safety attributable to 99mTc-ZHER2:41071 injections (ECG ) | 24 hours
  The safety attributable to 99mTc-ZHER2:41071 injections will be evaluated based on the assessments of ECG (% of cases with abnormal findings relative to baseline)
Safety attributable to 99mTc-ZHER2:41071 injections (blood laboratory tests) | 24 hours
  The safety attributable to 99mTc-ZHER2:41071 injections will be evaluated based on the blood laboratory tests (% of cases with abnormal findings relative to baseline)
Safety attributable to 99mTc-ZHER2:41071 injections (urine laboratory tests) | 24 hours
  The safety attributable to 99mTc-ZHER2:41071 injections will be evaluated based on the urine laboratory tests (% of cases with abnormal findings relative to baseline)
Safety attributable to 99mTc-ZHER2:41071 injections (incidence and severity of adverse events) | 24 hours
  The safety attributable to 99mTc- ZHER2:41071 injections will be evaluated based on the rate of adverse events (%)
Safety attributable 99mTc-ZHER2:41071 injections (concomitant medication) | 24 hours
  The safety attributable to 99mTc-ZHER2:41071 injections will be evaluated based on the rate of administration of concomitant medication (%)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Chernov, MD, Prof., Principal Investigator — Tomsk NRMC
Locations (1):
- TomskNRMC, Tomsk, Russia